

# INFORMATION ABOUT A UNIVERSITY OF WASHINGTON RESEARCH STUDY

#### The Asthma, Airport, and Air Pollution (AAA) Intervention Study

#### What is this study about?

We are conducting this study because we want to find out whether indoor air filtration can improve air quality and reduce asthma symptoms for children with asthma living near Seattle-Tacoma (Sea-Tac) International airport. When planes take off and land, they generate certain types of air pollution that might cause health problems for children with asthma. We aim to test different types of indoor air filters for effectiveness in reducing health risks of outdoor and indoor air pollution.

# Why are we asking you to be part of this study?

We are inviting you and your child to participate because you were referred to the King County Asthma Program. Our research team will work closely with the Asthma Program to coordinate your activities in this research study, if you choose to join, with you and your child's participation Asthma Program.

#### What will you be asked to do?

If you decide to be in this study, we will ask you to take part in a few study activities, listed in the table below. You, as the child's caregiver, will be the primary participant in these activities. Your child's involvement will be minimal. Study activities will begin soon after you enroll and last for about four months. Toward the end of your involvement in our research study, your child will begin the standard King County Asthma Program that you were referred to. Deciding to partipate in this study delays your child starting the Asthma Program by 3-4 months.

There will be two groups of participants, and the type of air filter put in your home will be based on your group. Your group assignment will be random, like the flip of a coin. There is a chance that the group you are assigned to does not improve air quality or asthma symptoms. We aim to enroll about 100 families in the study.

#### **PROCEDURES**

**Enrollment survey** – After you enroll, we will email you a link to an online survey. Topics will include basic demographics, your child's health history and current asthma health, your child's sleep, family health and health-related habits, and characteristics of your home. We will ask you to talk to your child about their recent asthma symptoms and medication use to answer a few of these questions. This survey should take less than 15 minutes to complete. You may also do this as part of Home Visit #1.



**Home visit #1** – The study team will visit your home sometime in the next month. You, the caregiver, should be at this home visit but your child does not need to attend. We will set up the air cleaner in your child's bedroom and an air pollution monitor. A team member will work with you to demonstrate and test out the text-based surveys you will receive over the next three months (see below.) You will receive partial compensation for your study participation at this time. The visit is expected to take about 30 minutes.

**Use of indoor air cleaner** – We will ask you to keep the air cleaner in your child's bedroom turned on whenever the child is at home. If you have any concerns or problems with this unit, you may call or email the study team.

Weekly surveys by text about your child's symptoms – For three months, you will receive texts every week with a few questions about your child's recent asthma symptoms and medication. It should take less than 5 minutes to respond to all the questions by text each time. If you do not respond that day, we will send you a reminder the next day. At the second home visit, you'll receive compensation for the number of weekly surveys completed.

**End of study survey** – You will complete a second online survey similar to the enrollment survey after you complete our study. In addition to some topics covered in the first survey, you will be asked about your experience in the study, including how you feel about the air cleaner that you used during the study. You may complete this survey online or at the time of Home Visit #2. This survey will be shorter than the first and take 5-10 minutes to complete.

**Home visit #2** – At the end of the study, the team will visit your home again to collect the air sensor. You will receive the remaining compensation for your participation as well as a new high-quality air filter. You will be allowed to keep the air cleaner. The visit is expected to take less than? 30 minutes.

#### Why might you want, or not want, to participate?

These are some reasons you may want to be in our study:

- We will provide an air cleaner for you to use during the study. Depending on your group assignment, you will receive one of two types of cleaners. One group will receive an air cleaner that may improve air quality and asthma symptoms and the other group will receive an air cleaner with a filter that may not improve air quality and asthma symptoms. At the end of the study, everyone in both groups will get to keep the air cleaner and will be given a high-efficiency filter to keep.
- We will measure indoor air pollution in your home for three months, and share the information collected with the Asthma Program team. It is possible that we learn about air pollution in your home specifically and the effectiveness of the air cleaner in decreasing air pollution in your home. This information may help the Asthma Program team provide better assistance to your family, improving the indoor environment and reducing triggers of asthma symptoms.
- You will receive compensation for your time and efforts, as described below.

Approved 2/22/2024 UW IRB.

W IRB These are also some reasons why you may not want to participate:

- If you enroll in this research study, your child will not begin the King County Asthma Program immediately. Instead, they will begin after a delay of three to four months. If your child has severe asthma, we will recommend that you begin the asthma program immediately and do not participate in research. To determine if this is the case, we will review information about your child's current asthma symptoms collected at the start of the study in collaboration with a pediatrician. Even if your child's asthma is not severe, you may prefer to skip this research opportunity so you can begin the Asthma Program sooner.
- Possible sleep disturbance due to the noise from the air cleaner.
- Safety precautions must be taken when using the air cleaner to avoid injury. For example: no playing
  with or climbing on the unit, no objects can be inserted into the vents, no touching the unit with wet
  hands, keep water away, and do not use near hot objects. Please see the <u>user manual</u> for a full list of
  safety precautions.
- Some spaces may not be suitable to fit the 15"(W) x 8.2" (D) x 23.6 in (H). You may not be able to participate if a suitable location or power source cannot be identified. There might be a small increase in the electric bill, running the filter at high power is of similar energy cost to keeping one 75W light bulb on for the duration of the study
- We will collect some information that identifies you and your child, including your names, phone
  number, and home address. We will keep this information secure, as described below, but there is still a
  possibility that study data are accidentally released.
- The research team will visit your home. They will be professional and respect your privacy and personal space. In addition, all study staff will have recent background checks and be trained to interact with children in a safe maner. However, it may be feel uncomfortable to have people you do not know in your home.
- The alternatives to participation is to start the PHSKC Asthma Program and to purchase a HEPA air filtration unit.

## How will we protect the information you provide?

We will protect your confidentiality. We will store your name and other identifiable information separate from the study data. Access to your identifying information will be limited to certain members of the study team and any individuals from the UW or other agencies that may need to audit study records. When we publish the

Approved 2/22/2024

results of this study, we will not use your name. Information about the study and your study results may be shared with the King County Asthma Program, because it may help them provide assistance to you and your child on how best to manage their asthma.

The information that we obtain from you for this study might be used for future studies. We may remove anything that might identify you from the information, including your home address, phone number, and names of you and your child. If we do so, the information may then be used without getting additional permission from you. If this future research does involve information that identifies you, a review board will decide whether or not we need to get additional permission from you.

What if you want to stop being in this study, or if the researcher decides you should no longer participate?

You may stop participation in this study at any point, for any reason. You may be withdrawn from the study and referred to care if you develop severe asthma as indicated by the weekly caregiver surveys. If you are withdrawn, you will keep the air cleaner with HEPA filters.

### Other information about this study.

**Being in this study is voluntary.** This means that you can refuse to sign up. It also means that if you do sign up, you can decide to stop being in the study at any time without penalty.

If you choose not to participate or you start but then choose to stop being in the study at any point, it will not affect your eligibility for the King County Asthma Program.

We are receiving financial support from the Washington State Department of Health to complete this study.

You will receive financial compensation for your time. All participants will be paid up to \$135, including \$50 delivered by gift card at the time of the first home visit. At the second home visit, you will receive an additional \$25 plus \$5 for each weekly asthma symptom survey completed during the study (up to \$60). As described above, you will also get to keep the HEPA air cleaner and replacement filters.

A copy of the consent form will be emailed to you at an email address that you provide. It will be a "PDF" document. Most computers already have PDF viewer software installed, which will allow you to open, read, or print the consent form. The email we send you will include a link to PDF viewer software (such as Adobe Acrobat



W IRB Reader) in case your computer doesn't already have it. If you would prefer to receive a paper copy of the consent form at no cost to you, please contact the researcher(s) listed in this consent form.

### What can you do if you want more information?

**Talk to the study team**. We are here to help you understand the study. Please ask us any questions you may have, even about things that are not in this document. It is our responsibility to give you the information you need to make a decision and to give you time to think about whether or not you want to sign up. If you feel you have been harmed by participating, you can contact us about that too.

**Talk to someone else**. If you want to talk about the study with someone who is not part of the study team, talk about your rights as a research subject, or to report problems or complaints about the study, contact the UW Human Subjects Division.

| Study Team | Maria Tchong French, Study Coordinator |
|----------------------------|------------------------------------------|
| | mitchong@uw.edu |
| | UW AAA Research Staff, General Questions |
| | <u>uwaaa@uw.edu</u> |
| UW Human Subjects Division | 206.543.0098 |
| | hsdinfo@uw.edu |

Printed name of study staff obtaining consent

Date

#### Subject's statement

By signing this consent form, I confirm that the study has been explained to me and I volunteer to participate in the research. I have had a chance to ask questions. If I have questions later about the research or feel I have been harmed by participating in the study, I can contact a member of the research team or the UW Human Subjects Division using the information listed above. I will receive a copy of this consent form.

Printed name of subject Signature of subject Date

Approved 2/22/2024 UW IRB

Document Date & Version 06.01.2023 posted

[AAA Consent]